CLINICAL TRIAL: NCT02507219
Title: Placebo-controlled, Dose-response Study of Ibuprofen Effects on Brain Function
Brief Title: Study of Ibuprofen Effects on Brain Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015-007-00
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive one dose of placebo (sugar pill) at one of the three testing sessions . Placebo capsules will be produced in the same manner as the ibuprofen by a local compounding pharmacy in Tulsa, OK.
  Interventions: Drug: Ibuprofen
- Ibuprofen, 200mg (Active Comparator): Subjects will receive one oral dose of 200mg at one of the three testing sessions. Ibuprofen capsules will be produced by a local compounding pharmacy in Tulsa, OK.
  Interventions: Drug: Ibuprofen
- Ibuprofen, 600mg (Active Comparator): Subjects will receive one oral dose of 600mg at one of the three testing sessions. Ibuprofen capsules will be produced by a local compounding pharmacy in Tulsa, OK.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — On the day of sessions 2-4, subjects will receive either placebo, 200 mg of ibuprofen or 600 mg of ibuprofen after signing the consent form for this study in a randomized, double-blind, counter balanced order. Each study session will occur 1-2 weeks following the previous session. Ibuprofen will be capsuled, and identical placebo capsules will be produced.
  Other Names: Placebo

SUMMARY:
The aim of this project is to determine whether the acute oral administration of Ibuprofen changes the activation pattern in the amygdala and other brain structures during functional magnetic resonance imaging. The investigators use a double-blind, randomized, repeated-measures design. Each of the 20 healthy control subjects will be tested three times and receive placebo, 200 mg or 600 mg dose of ibuprofen p.o. The study will consist of 4 sessions: a baseline screening session and 3 testing sessions scheduled 1-2 weeks apart. Each of these individuals will undergo a multi-level assessment based on the RDoC approach that consists of (a) a standardized diagnostic assessment, (b) self-report questionnaires assessing the positive and negative valence domains as well as interoception, (c) behavioral tasks assessing reward-related processing, avoidance, and aversive processing, cognition, and interoception; (d) physiological measurements consisting of facial emotion expression monitoring, heart rate and respiration, (e) functional magnetic resonance imaging focusing on reward-related processing, fear conditioning and extinction, cognitive inhibition, and interoceptive processing, and (f) biomarker assessments.

DETAILED DESCRIPTION:
Occasional OTC nonsteroidal anti-inflammatory drugs (NSAID) use is prevalent in the United States (25% aspirin, 9% ibuprofen, and 2% naproxen). An estimated 36 million Americans use over-the-counter (OTC) analgesics daily, however, considering the widespread use of analgesic agents, the overall incidence of serious drug-drug interactions involving these agents has been relatively low. Neuroinflammatory mechanisms have been implicated in depression, and NSAIDs have been found effective in animal models of depression both in monotherapy and when used to augment antidepressant drugs. However, results with NSAIDs have been mixed in human observational studies, with both better and worse depression outcomes reported. In animal studies, mice injected with BCG showed an increase in the total immobility time during the forced swim test (FST) and the tail suspension test (TST) and an increase in cerebral PGE2 and NO levels. Ibuprofen decreased the total immobility time during FST and TST and decreased cerebral PGE2 and NO levels, which was comparable to fluoxetine's effect. This would suggest that ibuprofen might have an antidepressant effect through inhibition of PGE2 and NO production.

Some studies have demonstrated the success of augmentation of antidepressant therapy with nonsteroidal anti-inflammatory drugs (NSAID) in decreasing depressive symptoms. However, little is known about the benefit of NSAID therapy on depressive symptoms. In a recent meta-analysis, using multivariable regression analysis a detectable effect in lowering PHQ-9 score in the ibuprofen or naproxen group (-0.31) and Celebrex group (-0.61) (p= .0390) was observed. However, in a study with cognitively normal volunteers age 70 and older with a family history of Alzheimer-like dementia who were randomly assigned to receive celecoxib 200 mg twice daily, naproxen sodium 220 mg twice daily, or placebo the investigators found no treatment effect on geriatric depression scores over time in the subgroup of participants with significant depressive symptoms at baseline. Moreover, there is some concern that anti-inflammatory drugs inhibit the antidepressant effects of SSRIs. In the only published fMRI study, ten healthy subjects underwent a double-blind, placebo-controlled, randomized, cross-over phFMRI study with somatosensory painful stimulation of the right median nerve. These authors reported a task-related increase of BOLD signal between drug and placebo in the primary somatosensory area and the middle frontal gyrus that was not related to changes in subjective pain scores. Thus there is some evidence that ibuprofen influences the BOLD response in specific pain-related brain areas. Taken together, there is mixed evidence for the effect of ibuprofen on mood and no data on its effect on the emotion circuitry.

Hypotheses:

1. The activation pattern in the amygdala during risk-taking decision-making will be attenuated by ibuprofen in a dose dependent manner.
2. The activation pattern in the amygdala during anticipatory emotional arousal will be attenuated by ibuprofen in a dose dependent manner.
3. The activation pattern in the amygdala during emotional face processing will be attenuated by ibuprofen in a dose dependent manner.
4. The behavioral response during tasks assessing emotional and cognitive processes including positive and negative valence and reward based learning will be modulated by ibuprofen in a dose dependent manner.

ELIGIBILITY:
Inclusion Criteria:

1. Male, or female
2. Between the ages of 18-50.
3. In good general health

Exclusion Criteria:

1. Subjects who report a history of any mental health disorder such as dysthymia, simple phobia, major depression, obsessive compulsive disorder or panic disorder as a primary diagnosis currently or within 6 months prior to the screening visit.
2. Subjects with a history of schizophrenia, schizoaffective disorder, or a bipolar disorder.
3. Subjects who report DSM-V criteria for substance use disorder (alcohol or drugs) currently or within 6 months prior to screening
4. Subjects who have a positive urine illicit drug screen.
5. Subjects that regularly (more than 15 days for past 30 days) use NSAIDS and have not used NSAIDS in the previous 5 days.
6. Subjects with a history of clinically significant hepatic cardiac, renal, neurologic, cerebrovascular, metabolic or pulmonary disease, gastric disease.
7. Subjects who have taken psychotropic drugs or antidepressants (including monoamine oxidase inhibitors, MAOI's) within the last year
8. Subjects with a history of seizure disorders (except for febrile seizures in childhood).
9. Subjects who, in the investigator's judgment pose a current, serious suicidal or homicidal risk or have made a suicide attempt within the past 6 months.
10. Women who have a positive serum HCG pregnancy test at screen visit or who are lactating or planning to become pregnant within the next 18 weeks following the screen visit.
11. Women who are currently menstruating.
12. The subject suffers from claustrophobia, or phobia for injections or blood.
13. Magnetic Resonance Imaging related exclusion criteria: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), subjects who have ever been a metal worker/welder; history of eye surgery/eyes washed out because of metal, aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, subjects who are in the first trimester of pregnancy, subjects with an I.U.D. (birth control device), a shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Paulus, M.D., Study Director — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Delaney JA, Biggs ML, Kronmal RA, Psaty BM. Demographic, medical, and behavioral characteristics associated with over the counter non-steroidal anti-inflammatory drug use in a population-based cohort: results from the Multi-Ethnic Study of Atherosclerosis. Pharmacoepidemiol Drug Saf. 2011 Jan;20(1):83-9. doi: 10.1002/pds.2065. Epub 2010 Nov 11. PMID 21182156
- [Background] Hersh EV, Pinto A, Moore PA. Adverse drug interactions involving common prescription and over-the-counter analgesic agents. Clin Ther. 2007;29 Suppl:2477-97. doi: 10.1016/j.clinthera.2007.12.003. PMID 18164916
- [Background] Andrade C. Antidepressant augmentation with anti-inflammatory agents. J Clin Psychiatry. 2014 Sep;75(9):975-7. doi: 10.4088/JCP.14f09432. PMID 25295422
- [Background] Saleh LA, Hamza M, El Gayar NH, Abd El-Samad AA, Nasr EA, Masoud SI. Ibuprofen suppresses depressive like behavior induced by BCG inoculation in mice: role of nitric oxide and prostaglandin. Pharmacol Biochem Behav. 2014 Oct;125:29-39. doi: 10.1016/j.pbb.2014.07.013. Epub 2014 Aug 4. PMID 25101545
- [Background] Iyengar RL, Gandhi S, Aneja A, Thorpe K, Razzouk L, Greenberg J, Mosovich S, Farkouh ME. NSAIDs are associated with lower depression scores in patients with osteoarthritis. Am J Med. 2013 Nov;126(11):1017.e11-8. doi: 10.1016/j.amjmed.2013.02.037. Epub 2013 Aug 29. PMID 23993259
- [Background] Fields C, Drye L, Vaidya V, Lyketsos C; ADAPT Research Group. Celecoxib or naproxen treatment does not benefit depressive symptoms in persons age 70 and older: findings from a randomized controlled trial. Am J Geriatr Psychiatry. 2012 Jun;20(6):505-13. doi: 10.1097/JGP.0b013e318227f4da. PMID 21775876
- [Background] Warner-Schmidt JL, Vanover KE, Chen EY, Marshall JJ, Greengard P. Antidepressant effects of selective serotonin reuptake inhibitors (SSRIs) are attenuated by antiinflammatory drugs in mice and humans. Proc Natl Acad Sci U S A. 2011 May 31;108(22):9262-7. doi: 10.1073/pnas.1104836108. Epub 2011 Apr 25. PMID 21518864
- [Background] Delli Pizzi S, Mantini D, Ferretti A, Caulo M, Salerio I, Romani GL, Del Gratta C, Tartaro A. Pharmacological functional MRI assessment of the effect of ibuprofen-arginine in painful conditions. Int J Immunopathol Pharmacol. 2010 Jul-Sep;23(3):927-35. doi: 10.1177/039463201002300329. PMID 20943065
- [Derived] Le TT, Kuplicki R, Yeh HW, Aupperle RL, Khalsa SS, Simmons WK, Paulus MP. Effect of Ibuprofen on BrainAGE: A Randomized, Placebo-Controlled, Dose-Response Exploratory Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Oct;3(10):836-843. doi: 10.1016/j.bpsc.2018.05.002. Epub 2018 Jun 23. PMID 29941380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants were recruited for the study at the Laureate Institute for Brain Research in Tulsa, Oklahoma.
Pre-assignment Details: 22 of 24 participants who signed informed consent were randomized. 2 participants withdrew from the study prior to randomization due to work schedule and no response to scheduling attempts.
Groups:
- Placebo, Ibuprofen 200mg, Ibuprofen 600mg: Subjects will receive one dose of placebo or ibuprofen at three testing sessions in a randomized, double-blind, counter-balanced order. In this arm, the subject will receive the doses in the following order: Placebo, Ibuprofen 200mg, Ibuprofen 600mg. Each study session will occur 1-2 weeks following the previous session. Ibuprofen will be capsuled, and identical placebo capsules will be produced.
- Placebo, Ibuprofen, 600mg, Ibuprofen 200mg: Subjects will receive one dose of placebo or ibuprofen at three testing sessions in a randomized, double-blind, counter-balanced order. In this arm, the subject will receive the doses in the following order: Placebo, Ibuprofen 600mg, Ibuprofen 200mg. Each study session will occur 1-2 weeks following the previous session. Ibuprofen will be capsuled, and identical placebo capsules will be produced.
- Ibuprofen, 200mg, Placebo, Ibuprofen 600mg: Subjects will receive one dose of placebo or ibuprofen at three testing sessions in a randomized, double-blind, counter-balanced order. In this arm, the subject will receive the doses in the following order: Ibuprofen 200mg, Placebo, Ibuprofen 600mg. Each study session will occur 1-2 weeks following the previous session. Ibuprofen will be capsuled, and identical placebo capsules will be produced.
- Ibuprofen 200mg, Ibuprofen 600mg, Placebo: Subjects will receive one dose of placebo or ibuprofen at three testing sessions in a randomized, double-blind, counter-balanced order. In this arm, the subject will receive the doses in the following order: Ibuprofen 200mg, Ibuprofen 600mg, Placebo. Each study session will occur 1-2 weeks following the previous session. Ibuprofen will be capsuled, and identical placebo capsules will be produced.
- Ibuprofen 600mg, Placebo, Ibuprofen 200mg; Ibuprofen 600mg, Ibuprofen 200mg, Placebo: Subjects will receive one dose of placebo or ibuprofen at three testing sessions in a randomized, double-blind, counter-balanced order. In this arm, the subject will receive the doses in the following order: Ibuprofen 600mg, Placebo, Ibuprofen 200mg. Each study session will occur 1-2 weeks following the previous session. Ibuprofen will be capsuled, and identical placebo capsules will be produced.
Period: Overall Study
Arm/Group | Placebo, Ibuprofen 200mg, Ibuprofen 600mg | Placebo, Ibuprofen, 600mg, Ibuprofen 200mg | Ibuprofen, 200mg, Placebo, Ibuprofen 600mg | Ibuprofen 200mg, Ibuprofen 600mg, Placebo | Ibuprofen 600mg, Placebo, Ibuprofen 200mg | Ibuprofen 600mg, Ibuprofen 200mg, Placebo
Started | 5 | 4 | 3 | 3 | 4 | 3
Completed | 4 | 4 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is based on the 20 participants who completed all 3 arms of the study: placebo, ibuprofen 200mg and 600mg. The 2 participants who entered drug randomization but did not complete the study are not included. The 2 participants who signed informed consent but were not randomized are also not included.
Groups:
- All Study Participants: Subjects received either placebo, 200 mg of ibuprofen or 600 mg of ibuprofen after signing the consent form for this study in a randomized, double-blind, counter-balanced study. Each participant received all interventions. Each study session occurred 1-2 weeks following the previous session. Ibuprofen was capsuled, and identical placebo capsules were produced.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.75 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Dose-dependent Differences in the BOLD Response to fMRI Tasks in the Amygdala
Description: Change in amygdala activation following administration of placebo, 200mg of ibuprofen or 600mg of ibuprofen
Time Frame: 3-6 weeks
Population: Scans that had average Euclidean norm of motion parameters less than 0.15 were included in the analyses.
Measure: Mean (Standard Error); unit: percent signal change
Arm/Group | Placebo | Ibuprofen, 200mg | Ibuprofen, 600mg
Number analyzed (Participants) | 19 | 18 | 19
percent signal change
  Left amygdala | 0.20 (0.045) | 0.21 (0.032) | 0.23 (0.047)
  Right amygdala | 0.23 (0.037) | 0.23 (0.037) | 0.17 (0.063)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen, 200mg vs Ibuprofen, 600mg; A linear mixed effects model was run for the left amygdala with contrast and percent signal change between faces and shapes as the dependent variable and ibuprofen dose as a continuous predictor. Each subject had up to 3 visits and each visit contained 3 contrasts (happy - shape, angry - shape, fearful - shape) so subject and drug were used as random effects. Drug was nested inside of subject; Test type: Superiority; p = 0.512, Mixed Models Analysis; Slope = 0.000055, 95% CI 2-sided [-0.00011 to 0.00022] — Slope is percent signal change per milligram of ibuprofen
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen, 200mg vs Ibuprofen, 600mg; A linear mixed effects model was run for the right amygdala with contrast and percent signal change between faces and shapes as the dependent variable and ibuprofen dose as a continuous predictor. Each subject had up to 3 visits and each visit contained 3 contrasts (happy - shape, angry - shape, fearful - shape) so subject and drug were used as random effects. Drug was nested inside of subject; Test type: Superiority; p = 0.221, Mixed Models Analysis; Slope = -0.00012, 95% CI 2-sided [-0.00030 to 0.000067] — Slope is the percent signal change per mg of ibuprofen

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen, 200mg | Ibuprofen, 600mg
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes